CLINICAL TRIAL: NCT03037892
Title: A Prospective Randomized Comparative Study to Evaluate the Use of Remifentanil as a Sole Agent or in Combination With Midazolam Versus Fentanyl/Midazolam During Sedation for Colonoscopy
Brief Title: Comparison of Remifentanil as a Sole Agent or in Combination With Midazolam Versus Fentanyl/Midazolam During Sedation for Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Hamad University Hospital, Bahrain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KHUH/Research/No.89/2015
Record Dates: First submitted 2015-08-24; First posted 2017-01-31 (Estimated); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: Colonoscopy
MeSH Terms: interventions — Midazolam; Fentanyl; Remifentanil

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Midazolam and Fentanyl (Active Comparator): Midazolam and Fentanyl Two minutes before the colonoscopy procedure, a bolus of midazolam 0.03mg/Kg and 1.5microgram/Kg fentanyl will be given intravenously over 60 sec in group 1. 0.5 mg of midazolam intravenously can be given every two minutes till the patient is sufficiently sedated (sleeping but arousable on calling). The colonoscopy can start at this end point. Increments of 0.5mcg/Kg of fentanyl will be given if patient complains of pain, which can be repeated every 5 minutes if there is persistent pain
  Interventions: Drug: Midazolam, Fentanyl
- Midazolam and Remifentanil (Experimental): Midazolam and Remifentanil Target controlled infusion of Remifentanil to 3.0 ng/ml will be started 2 minutes before procedure. The patient will then be given same doses of midazolam in 0.5 mg increments till sedated sufficiently (sleeping but arousable on verbal command). During Colonoscopy the dose of Remifentanil could be increased by 0.5ng/ml if patient complained of pain upto 4.0ng/ml.
  Interventions: Drug: Midazolam, Remifentanil
- Remifentanil (Experimental): Remifentanil Group Patients will receive only Remifentanil in the same doses as given in group 2. During the procedure if the pain is excessive and persistent in spite of increasing the respective doses as prescribed in each group, or causing loss of cooperation of patient and interfering in the performance of procedure, the patients will be given sleep dose of Inj Propofol and further anaesthesia care as required will be provided for same.
  Interventions: Drug: Remifentanil

INTERVENTIONS:
Drug: Midazolam, Fentanyl — Two minutes before the colonoscopy procedure, a bolus of midazolam 0.03mg/Kg and 1.5microgram/Kg fentanyl will be given intravenously over 60 sec in group 1. 0.5 mg of midazolam intravenously can be given every two minutes till the patient is sufficiently sedated (sleeping but arousable on calling). The colonoscopy can start at this end point. Increments of 0.5mcg/Kg of fentanyl will be given if patient complains of pain, which can be repeated every 5 minutes if there is persistent pain.
  Arms: Midazolam and Fentanyl
Drug: Midazolam, Remifentanil — The patient in group 2 Target controlled infusion of Remifentanil to 3.0 ng/ml will be started 2 minutes before procedure. The patient will then be given same doses of midazolam in 0.5 mg increments till sedated sufficiently (sleeping but arousable on verbal command). During Colonoscopy the dose of Remifentanil could be increased by 0.5ng/ml if patient complained of pain upto 4.0ng/ml.
  Arms: Midazolam and Remifentanil
Drug: Remifentanil — The group 3 patient will receive only Remifentanil in the same doses as given in group
  Arms: Remifentanil

SUMMARY:
Colonoscopy is one of the most commonly performed outpatient procedure for diagnosis and treatment of lower gastrointestinal tract disorders. It has been largely accepted as an effective tool for colorectal cancer(CRC) screening, given its ability to detect and remove identified polyps. Increased colonoscopy utilization is associated with the observed decline in the incidence of CRC and its diagnosis at earlier stages. Diagnostic and therapeutic colonoscopy can successfully be performed using moderate sedation in the ambulatory setting. Techniques of sedation must guarantee the comfort and safety of patients, and at the same time allow a rapid turnover of patients.. An anaesthetic agent with rapid onset and offset of action, and convenient titration of anaesthetic/analgesic depth as well as rapid recovery to enable discharge from the endoscopy unit as soon as possible would be ideal as most such procedures are performed in the Non-Operating Room Anaesthesia(NORA) settings.

There is recent interest in the use of Remifentanil, in endoscopic units as it might have advantages over other drugs because of its profound analgesic effects, rapid onset and offset time and rapid titration to the individual patient's requirements and intermittent pain during colonoscopy.

The aim of this randomized study is to test the hypothesis that a colonoscopy of good quality in terms of pain relief, patient comfort and discharge times with less cardiorespiratory side effects can be performed using Remifentanil as a sole agent as compared with the standard midazolam/fentanyl protocol. The second group combining Remifentanil with Midazolam is taken to evaluate if there is any advantage of adding an anxiolytic amnesic drug as used in the standard Midazolam/Fentanyl Protocol.

DETAILED DESCRIPTION:
A Prospective Randomized Comparative Study to Evaluate the Use of Remifentanil as a Sole Agent or in Combination with Midazolam Versus Fentanyl/Midazolam during Sedation for Colonoscopy.

Background:

Audits of patient experiences and studies on quality improvement for colonoscopy have shown that increased sedation administration results in long-lasting improvement of colonoscopy quality indicators. However deep sedation in NORA ambulatory settings has been associated with increased sedation associated risks and raises costs for healthcare providers. Sedation may delay discharge of patients or cause discharge of patients with early cognitive impairment that contraindicate complex activities of daily living, The search is still on for an ideal drug that produces optimal operating conditions with minimum postoperative cognitive impairment.

Remifentanil is an ultrashort, very potent narcotic, which is eliminated by plasma and tissue esterases. There is recent interest in the use of Remifentanil in endoscopic units as it might have advantages over other drugs because of its profound analgesic effects, rapid onset and offset time and rapid titration to the individual patient's requirements and intermittent pain during colonoscopy. There are a few studies which suggest that the analgosedation(intense pain relief without loss of consciousness) achievable with remifentanil is a valid alternative to the present sedo-analgesia techniques used for colonoscopic sedation.

Ackcaboy ZN conducted a prospective randomized trial to test the hypothesis that continuous infusion of low dose remifentanil (0.05mcg/kg/min) continuous and bolus injection - in combination with 2 mg of midazolam, can provide effective analgesia, sedation, amnesia, patient comfort and stable recovery profile without respiratory depression when compared with Propofol infusion during colonoscopy.

Following Moerman's hypothesis: "If pain is the crucial point, why do we need sedation?", the use of remifentanil as a sole agent for colonoscopy, has been investigated and compared with the sedative scheme of midazolam plus pethidine. Remifentanil was found to provide sufficient pain relief with better hemodynamic stability, less respiratory depression, and significantly faster recovery and hospital discharge than moderate sedation with midazolam and pethidine. Midazolam-Fentanyl and Midazolam-Remifentanyl techniques has been compared for Endoscopic Retrograde Cholangio- Pancreatography another painful endoscopic procedure and there were definite advantages seen in the midazolam-remifentanil group in level of sedation and patient satisfaction. However, remifentanil use is not widespread and is being used only by anaesthesiologists.

There is scope to conduct further studies to ascertain if there is an actual real benefit of using remifentanil as a sole agent or in combination with midazolam, over the standard technique of midazolam/fentanyl used in endoscopy units.

This Controlled Randomized Clinical Study is planned to evaluate whether Remifentanil by itself as a sole agent or in combination with Midazolam provides a safe and effective sedation for colonoscopy as compared to the present technique of midazolam and fentanyl being used by most endoscopists.

1. Statement of the problem Colonoscopy is a proven method for bowel cancer screening and is often experienced as a painful procedure. They are the most frequently performed endoscopic procedures. However motivating patients to participate in colonoscopy screening continues to be a challenge as it is associated with considerable anxiety and pain. Additionally patients complain of disruption of normal activities by bowel preparations and hangover effects from sedation and need for an escort after procedure. The sedation protocol are followed by the endoscopists' themselves with a nurse who is monitoring the case. Rescue from extreme sedation or agitation is not uncommon. Ideal sedation should be potent and easily titrated , be adequate and safe for the painful procedure yet have a quick recovery for an early discharge as these procedures are usually done in an ambulatory setting.

Remifentanyl is a relatively new drug which has been used in endoscopic suites with some advantage. There is scope to conduct further studies to ascertain if there is an actual real benefit of using remifentanil as a sole agent or in combination with midazolam, over the standard technique of midazolam/fentanyl..

Significance of the problem

Colonoscopy is one of the most commonly performed outpatient procedure for diagnosis and treatment of lower gastrointestinal tract disorders, usually performed under moderate sedation in the ambulatory setting. As pain and vasovagal reactions are common during the procedure, administration of sedation and analgesia is imperative. Techniques of sedation must guarantee the comfort and safety of patients, and at the same time allow a rapid turnover of patients. An anaesthetic agent with rapid onset and offset of action, and convenient titration of anaesthetic/analgesic depth as well as rapid recovery to enable discharge from the endoscopy unit as soon as possible would be ideal.

There is recent interest in the use of Remifentanil in endoscopic units as it might have advantages over other drugs because of its profound analgesic effects, rapid onset and offset time and rapid titration to the individual patient's requirements and intermittent pain during colonoscopy. Remifentanil was found to provide sufficient pain relief with better hemodynamic stability, less respiratory depression, and significantly faster recovery and hospital discharge than moderate sedation in a few preliminary studies.

Objectives of the study:

General objective:

The study plans to study whether Remifentanil by itself as a sole agent or in combination with Midazolam provides a safe and effective sedation for colonoscopy as compared to the present technique of midazolam and fentanyl being used by the endoscopists.

Specific objective:

* Whether remifentanyl as a sole agent was effective and safe for Colonoscopies, or if combined with midazolam offered any advantages over the only remifentanyl or standard midazolam fentanyl technique.
* Effectiveness will be judged by the number of patients who complained of pain during procedure, number of patients who became uncooperative during the technique and had to be given Propofol to convert it into a general anaesthetic.
* Safety will be judged by any significant haemodynamic or respiratory changes and changes in sedation level in the various study groups.
* Advantages in reduced recovery time will be noted from the time to full recovery after sedation procedure.
* Patient and Endoscopist's satisfaction score will be recorded to see any differences in the three groups.

Method:

Following an Ethics Committee approval, 90 patients who are undergoing colonoscopy under moderate sedation in an ambulatory setting at Awali Hospital will be included in the study who satisfy the inclusion/exclusion criteria. Informed Consent will be taken preoperatively and they will be randomly allocated in to three groups as follows:

Group 1 - Patients will receive Midazolam and Fentanyl.

Group 2 - Patients will receive Midazolam and Remifentanil

Group 3 - Patients will receive Remifentanil as a sole agent

Study subjects: Inclusion and exclusion criteria of the study subjects.

Design: Prospective, randomized controlled clinical trial

Sample size: 90 patients will be selected for the study randomly dividing them into the three groups of 30 each.

Sampling technique: All patients due for colonoscopy under moderate sedation who satisfy the inclusion and exclusion criteria and who agree to be part of the study group by an informed consent will be randomly divided into the three groups of 30 each.

Randomization will be done by making identical folded slips of the three groups and by randomly picking up a slip preoperatively on the morning of procedure for each patient.

Timeframe of the study. The study will be done prospectively once approved by the Ethics Committee and registered as a Prospective Clinical Trial in the Registry

Data Collection methods, instruments used and measurements: Describe the instruments to be used for data collection (questionnaire, observation recording form, etc.)

Study Protocol:

Patients undergoing elective colonoscopy who satisfy the inclusion criteria will be randomly allocated to the 3 groups after taking an informed consent. All colonoscopies will be performed by two Endoscopists of Awali Hospital who seem to work in a very similar manner for colonic endoscopy.

On arrival to the endoscopy room an IV access will be established. Supplemental oxygen 3 L/min will be given through both the nostrils and mouth by a specially designed mask which can monitor the end tidal CO2 level. The basal values of noninvasive blood pressure (NIBP), peripheral oxygen saturation (SpO2), heart rate (HR), respiratory rate (RR) and end-tidal CO2 level (ETCO2) will be noted.

Two minutes before the colonoscopy procedure, a bolus of midazolam 0.03mg/Kg and 1.5microgram/Kg fentanyl will be given intravenously over 60 sec in group 1. 0.5 mg of midazolam intravenously can be given every two minutes till the patient is sufficiently sedated (sleeping but arousable on calling). The colonoscopy can start at this end point. Increments of 0.5mcg/Kg of fentanyl will be given if patient complains of pain, which can be repeated every 5 minutes if there is persistent pain. The patient in group 2 Target controlled infusion of Remifentanil to 3.0 ng/ml will be started 2 minutes before procedure. The patient will then be given same doses of midazolam in 0.5 mg increments till sedated sufficiently (sleeping but arousable on verbal command). During Colonoscopy the dose of Remifentanil could be increased by 0.5ng/ml if patient complained of pain upto 4.0ng/ml. The group 3 patient will receive only Remifentanil in the same doses as given in group 2. During the procedure if the pain is excessive and persistent in spite of increasing the respective doses as prescribed in each group, or causing loss of cooperation of patient and interfering in the performance of procedure, the patients will be given sleep dose of Inj Propofol and further anaesthesia care as required will be provided for same.

The Haemodynamic Parameters(NIBP,HR), RR, SPO2, Sedation Scare (Ramsay) and ETCO2 will be measured 1 and 3 min after the drug dose then every 5 min till end of procedure. After procedure the patients will be shifted to recovery and the same parameters will continue to be measured every 5 min until discharge from the 30 min stay in the recovery room. Pain Scoring will be done by a Visual Analog Pain Score (VAS) (0- minimum to 100mm- Maximum pain) just after passing the scope, during the scope, just after the completion of colonoscopy and at the discharge from the recovery unit.

Total amount of drug consumed, duration of colonoscopy, incidence of adverse effects (desaturation <94% on Pulseoximetry, Hypoventilation (RR<8/min or apneic episode, hypotension (SBP<90mm Hg), nausea vomiting or pruritis will be recorded.

Patient satisfaction will be noted at the time of discharge from ward

Primary Outcome Measures:

• The Recovery Time The patient will be considered recovered if and when they achieve an Aldrete score of 10. Aldrete scoring will be done every 5 minutes after completing colonoscopy up to 30 min or till achievement of a 10/10 Aldrete Score.

Aldrete score

* Respiration: Able to take deep breath and cough = 2, Dyspnea/shallow breathing = 1, Apnea = 0
* O2 saturation: Maintains > 92% on room air =2, Needs O2 inhalation to maintain O2 saturation > 90% =1 , O2 saturation < 90% even with supplemental oxygen =0
* Consciousness: Fully awake= 2, Arousable on calling = 1, Not responding = 0
* Circulation: BP +/- 20 mm Hg preop =2, BP +/- 20-50 mm Hg preop =1, BP +/- 50 mm Hg preop =0
* Activity: Able to move 4 extremities = 2, Able to move 2 extremities = 1, Able to move 0 extremities 0
* Participants Assumed to Feel Frequent Pain, during and after colonoscopy. • Patients sound "Ah" at feeling pain during colonoscopy would be taken as a measure: if a patients sounds "Ah" > 6 times, the patient was assumed to feel frequent pain. Will be scored as 0 no pain ,1if he complains of pain or 2 if he says Ah or complains of pain frequently, that is, more than 6 times.
* Patient's Distress Score every 5 min till the end of colonoscopy. Patients' distress as minimal, mild moderate or severe distress.
* Number of patients in each group who had to receive propofol due to loss of cooperation

Secondary Outcome Measures:

* Endoscopist Satisfaction. Time Frame: 5 min after the colonoscopy. Endoscopist's satisfaction after colonoscopy in visual analogue scale 100 mm
* Incidence of Patient's Recall. Tested after colonoscopy before discharge from the hospital. The numbers of patients who recalled instructions and explanations given during colonoscopy will be noted and if there was any unpleasantness related to the recall or awareness.
* Patient satisfaction. Will be tested on a numerical scale from 0 (not satisfied at all) to 10 (fully satisfied) at the time of discharge from the hospital.
* Side Effects noted in each group for example excessive sedation, nausea, vomiting, pruritis, respiratory depression or apnoea.

The data will be statistically analyzed, to arrive at a conclusion on whether remifentanyl as a sole agent was effective for Colonoscopies, or if combined with midazolam offered any advantages over the only remifentanyl or standard midazolam fentanyl technique.

Implications of the study results to population health and health system policy in Awali Hospital and Bahrain:

ELIGIBILITY:
Inclusion Criteria:

1. Patients between 18-75 years
2. ASA Grade I, II and controlled ASA III.

Exclusion Criteria:

1. Patient Refusal
2. Patients with psychiatric or Emotional Disorders
3. Previous adverse reaction to any of the drugs used
4. History of addiction to opiates/sedatives/alcohol
5. ASA Grade 3-4 patients with clinically significant or uncontrolled cardiovascular or respiratory disease.
6. Pregnancy
7. Age <=18years

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
The Recovery Time | 30 min
  Every 5 minutes till a score of 10/10 achieved on Aldrete Score
propofol consumption | 60 minutes
  Number of patients in each group who had to receive propofol due to loss of cooperation

SECONDARY OUTCOMES:
Endoscopist Satisfaction | 60 min
  Endoscopist Satisfaction scored from 1-10
Incidence of Patient's Recall. | 6 hours
  Any recall and unpleasantness related to recall will be noted
Patient satisfaction | 6 hours
  Patient satisfaction. Will be tested on a numerical scale from 0 (not satisfied at all) to 10 (fully satisfied) at the time of discharge from the hospital.
Side effects | 6 hours
  Side Effects noted in each group for example excessive sedation, nausea, vomiting, pruritis, respiratory depression or apnoea.

CONTACTS AND LOCATIONS:
Overall Officials: Reeta Singh, MD DNBE MBA, Principal Investigator — Awali Hospital
Locations (1):
- Awali Hospital, Manama, Bahrain